CLINICAL TRIAL: NCT06666608
Title: The Efficacy of Bone Stimulator in Treatment and Return-to-Sport for Spondylolysis
Brief Title: Bone Stimulator for Spondylolysis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Methodist Hospital Research Institute (Other)
Responsible Party: Principal Investigator, Mark Prasarn, Orthopedic Surgeon, The Methodist Hospital Research Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRO00038514
Record Dates: First submitted 2024-10-28; First posted 2024-10-30 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Spondylolysis; Symptomatic Spondylolysis; Athletes
MeSH Terms: conditions — Spondylolysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Bone Stimulator Treatment (Experimental): In addition to the standard of care treatment at Houston Methodist for spondylolysis (provision of a back brace and prescribed physical therapy regimen), participants assigned to this group will be provided a bone stimulator wherein they will be asked to wear their device for a minimum of 30 minutes a day for 12 weeks with no maximum usage time. The device will track compliance, and will be worn when at rest.
  Interventions: Device: Bone Stimulator
- Standard of Care Treatment (Active Comparator): Participants assigned to this group will undergo the standard of care treatment for spondylosis which is physical therapy and the usage of a back brace.
  Interventions: Other: Standard of Care Spondylolysis Treatment

INTERVENTIONS:
Device: Bone Stimulator — Subjects will be asked to wear their device (if applicable) for a minimum of 30 minutes a day for 12 weeks with no maximum usage time. The device will track compliance. Bone stimulator should be worn at rest.
  Arms: Bone Stimulator Treatment
Other: Standard of Care Spondylolysis Treatment — Participants will follow the standard of care regimen for spondylolysis treatment at Houston Methodist which will involve physical therapy and wearing a back brace.
  Arms: Standard of Care Treatment

SUMMARY:
This prospective study aims to investigate the effectiveness of bone stimulator therapy as adjunct treatment of spondylolysis in athletic populations. By evaluating its impact on pain reduction, functional improvement, osseous bony union and return-to-sport time, the investigators seek to provide valuable insights into the role of bone stimulation therapy as a potential treatment modality for this challenging condition.

ELIGIBILITY:
Inclusion Criteria:

* Patients between the ages of 16 to 40 years of age diagnosed with symptomatic spondylolysis by one of the investigators
* Patients who plan to attend prescribed physical therapy
* Patients who participate in a regular sport whether that be professional, collegiate or recreational

Exclusion Criteria:

* Any condition which in the investigator's opinion, would interfere with the subject's ability to comply with study instructions
* Patients with contraindications to bone stimulator therapy
* Patients with pacemaker and implantable cardioverter defibrillator
* Patients with previous spine surgery
* Patients with metabolic bone conditions
* Patients who use nicotine products
* Vulnerable populations
* Non-English speaking services

Ages: 16 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Time to Return to Sport After Diagnosis of Spondylolysis and Bone Healing | Baseline visit, 6 weeks after baseline, 12 weeks after baseline, 6 months after baseline
  This outcome will be evaluated via REDCap with a Return to Sport Questionnaire, which will ask what sport(s) participant played prior to injury, if they have returned to the sports they played prior to back injury, what level of sports they returned to (recreational, organized, professional), what level of play they have returned to (same as before injury, higher than before injury, or lower than before injury), and if they report that they did not return to sport, what the reason was. This outcome will also be evaluated by the Tegner Activity Level, which will ask participants to rate their highest level of activity they participated in before their injury and at the current moment on a scale of 0 to 10 where 0 is sick leave or disability pension because of spine problems and 10 is competitive sports at the national elite level.

SECONDARY OUTCOMES:
Level of pain | Baseline visit, 6 weeks after baseline, 12 weeks after baseline, 6 months after baseline
  Pain levels will be assessed with the visual analog scale, which asks patients to place a mark on a scale from no pain to worst possible pain level where they think their pain level is best represented.
Level of pain | Baseline visit, 6 weeks after baseline, 12 weeks after baseline, 6 months after baseline
  Pain levels will be assessed with one question on the Oswestry Disability Index which asks about a subjective rating of pain intensity from "I have no pain at the moment" to "the pain is the worst imaginable at the moment."
Effect on Daily Life | Baseline visit, 6 weeks after baseline, 12 weeks after baseline, 6 months after baseline
  This outcome will be measured with the Oswestry Disability Index which asks participants to rate various aspects of their lives with subjective measures on how they are faring with daily tasks such as personal care, lifting, walking, sitting, social life, travel, etc. This scale consists of ten questions which are each scored from 0 to 5. A higher total cumulative score reflects worse outcomes with 81-100% indicating a participant is bedbound, and lower scores indicating better outcomes with 0-20% reflecting little hindrance to ability to cope with daily life.

OTHER OUTCOMES:
Physical Therapy Attendance | Baseline visit, 6 weeks after baseline, 12 weeks after baseline, 6 months after baseline
  Attendance at physical therapy will be tracked through EPIC as part of study participation.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Prasarn, MD, Principal Investigator — The Methodist Hospital Research Institute
Locations (1):
- Houston Methodist Hospital, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No